CLINICAL TRIAL: NCT07253129
Title: Allogeneic Hematopoietic Stem Cell Transplantation Versus Autologous Hematopoietic Stem Cell Transplantation for Peripheral T-cell Lymphoma Patients With Partial Remission After First-line Systemic Therapy : A Prospective, Multicenter, Cohort Study(T-START-PR)
Brief Title: Allo-HSCT Vs. Auto-HSCT for PTCL Patients With PR After First-line Systemic Therapy : A Prospective, Multicenter, Cohort Study-(T-START-PR)
Acronym: T-START-PR
Status: Recruiting | Type: Observational
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: T-START-PR
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Peripheral T Cell Lymphoma
Keywords: peripheral T cell lymphoma; allogeneic hematopoietic stem cell transplantation; autologous hematopoietic stem cell transplantation; partial response
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Allo-HSCT: Allo-HSCT involves the infusion of stem cells collected from a donor (genetically similar, but not identical)
  Interventions: Procedure: Allogenic stem cell transplant (ASCT)
- Auto-HSCT: Auto-HSCT involves the infusion of the patient's own previously collected stem cells.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Auto-HSCT involves the infusion of the patient's own previously collected stem cells.
  Other Names: Auto-HSCT
  Groups: Auto-HSCT
Procedure: Allogenic stem cell transplant (ASCT) — ASCT involves the infusion of stem cells collected from a donor (genetically similar, but not identical).
  Other Names: ASCT; Allo-HSCT
  Groups: Allo-HSCT

SUMMARY:
This study is a multicenter, two-arm, prospective clinical trial, comprising two groups: the allogeneic hematopoietic stem cell transplantation group (Allo-HSCT) and the autologous hematopoietic stem cell transplantation group (Auto-HSCT). It aims to evaluate the efficacy and safety of Auto-HSCT and Allo-HSCT in the treatment of peripheral T-cell lymphoma that has achieved partial response (PR) after first-line therapy. During the screening/baseline period, informed consent will be obtained, and inclusion/exclusion criteria will be verified. Group assignment (Allo-HSCT vs. Auto-HSCT) will be determined taking into account the availability of a matched donor and the patient's preference. The study plans to enroll 44 patients in the allogeneic hematopoietic stem cell transplantation group, while all concurrent patients undergoing autologous stem cell transplantation will be included in the other group for inverse probability weighting analysis. Data on demographics and medical history will be collected, and assessments including vital signs, physical examination, PET-CT, bone marrow aspiration smear, flow cytometry, and bone marrow pathology will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Age & Sex:

   Males or females aged 18 to 70 years (inclusive).
2. ECOG performance status score of 0 to 1, with no deterioration within the last two weeks.
3. Expected survival period greater than 12 weeks.
4. Patients must have a histopathological confirmation of PTCL according to the 2016 revised WHO classification of lymphoid neoplasms (Swerdlow SH et al. 2016). Eligible histological subtypes are limited to the following:

   * Peripheral T-cell lymphoma, not otherwise specified (PTCL-NOS)
   * Anaplastic large cell lymphoma, ALK-negative (ALK-ALCL)
   * Follicular helper T-cell lymphoma or PTCL with TFH phenotype (FTCL or PTCL-TFH)

   Patients undergoing allogeneic hematopoietic stem cell transplantation must have a suitable stem cell donor:

   (i) Related donors must be at least 5/10 matched for HLA-A, -B, -C, -DQB1, and -DRB1.

   (ii) Unrelated donors must be at least 8/10 matched for HLA-A, -B, -C, -DQB1, and -DRB1.
5. Patients must have achieved a partial response (PR) as per the Lugano 2014 response criteria for lymphoma after six cycles of CHOP, BV-CHP or CHOP-like chemotherapy.
6. Hematopoietic Cell Transplantation-Comorbidity Index (HCT-CI) score ≤ 2.
7. Adequate hepatic, renal, cardiac, and pulmonary function, defined as follows:

   1. Hepatic function: Serum total bilirubin ≤ 2 × upper limit of normal (ULN) (≤ 3.0 × ULN in cases of Gilbert's syndrome or baseline hepatic involvement); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN (≤ 5.0 × ULN in cases of hepatic involvement).
   2. Renal function: Serum creatinine ≤ 1.5 × ULN, or creatinine clearance ≥ 50 mL/min as calculated or measured by the Cockcroft-Gault method.
   3. Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 50% as measured by multigated acquisition (MUGA) scan or echocardiography (ECHO).
   4. Baseline oxygen saturation > 92%.
   5. Pulmonary function: Diffusing capacity of the lung for carbon monoxide (DLCO) (hemoglobin-corrected) ≥ 40% and forced expiratory volume in 1 second (FEV1) ≥ 50%.

Exclusion Criteria:

1. Ann Arbor clinical stage I disease.
2. History of malignancy within the past 5 years, except for locally curable malignancies that have been treated with curative intent (e.g., basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast).
3. Active infection, including:

   1. Known active or latent tuberculosis, evidenced by a positive tuberculin (PPD) skin test (induration >10 mm or per local criteria for a positive result) or radiographic findings suggestive of active/latent TB on chest X-ray/CT.
   2. Known history of infection with Human Immunodeficiency Virus (HIV) and/or AIDS.
   3. Chronic active hepatitis B or hepatitis C infection:

   <!-- -->

   1. Patients positive for hepatitis B virus (HBV) DNA are excluded; however, those with undetectable HBV DNA levels are eligible. The upper limit of normal (ULN) for HBV DNA shall be based on the reference values of each participating center.
   2. Patients positive for hepatitis C virus (HCV) RNA are excluded; however, those with undetectable HCV RNA are eligible. The ULN for HCV RNA shall be based on the reference values of each participating center.

   (d) Active viral infections other than hepatitis B or hepatitis C (e.g., herpes zoster, cytomegalovirus).

   (e) Infection requiring intravenous antimicrobial therapy, associated with hemodynamic instability, worsening or new onset of infectious signs/symptoms, or new infectious foci on imaging; or persistent fever without localizing signs that cannot rule out infection.

   (f) Positive serum DNA test for Epstein-Barr virus (EBV).
4. Poorly controlled cardiac symptoms or disease, such as:

   i. Heart failure greater than New York Heart Association (NYHA) class II. ii. Unstable angina. iii. Myocardial infarction within the past year. iv. Clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention.
5. Pregnant or lactating women, and subjects of childbearing potential unwilling to use effective contraception.
6. Psychiatric illness or individuals unable to provide informed consent.
7. PTCL patients with central nervous system involvement.
8. PTCL patients who have previously received PD-1 inhibitor therapy.
9. Any other condition that, in the judgment of the investigator, would make the subject unsuitable for participation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PTCL who are in PR following first-line therapy and who are both medically eligible and willing to undergo transplantation will be directly assigned to treatment with either allogeneic PBSCT or autologous HSCT.
Sampling Method: Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2029-05-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
2y-event-free survival (EFS) | up to 2 years for the 2y-EFS
  2-year event-free survival (EFS) rates post-transplant. An event is defined as whichever of the following occurs first: disease progression, death from any cause, commencement of new anti-tumor therapy, or a treatment-related serious adverse event (specifically including disabling events or secondary neoplasms). Subjects who were event-free at the data cutoff will be censored on the date of their last tumor assessment.

SECONDARY OUTCOMES:
3m and 6m-complete response rate | up to 3 months for the 3m-CR and up to 6 months for the 6m-CR
  The duration from the date of hematopoietic stem cell transplantation to the first occurrence of complete response.
1y and 2y-cumulative relapse rates (CIR) | up to 1 years for the 1y-CIR and up to 2 years for the 2y-CIR
  The cumulative probability of disease progression (including relapse or progression of the primary disease) within 1 or 2 years after transplantation, with non-progression-related death treated as a competing event.
1y and 2y-overall survival (OS) | up to 1 years for the 1y-OS and up to 2 years for the 2y-OS
  The probability of survival at 1 or 2 years, measured from the date of transplantation to death from any cause. Patients who are still alive at the time of analysis will be censored on the last follow-up date.
non-relapse mortality (NRM) | up to 1 years
  Death occurring after transplantation due to causes other than disease relapse, such as infection, organ toxicity, or transplantation-related complications. Deaths from any cause in the absence of prior relapse are considered events for this endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmitz N, Truemper L, Bouabdallah K, Ziepert M, Leclerc M, Cartron G, Jaccard A, Reimer P, Wagner E, Wilhelm M, Sanhes L, Lamy T, de Leval L, Rosenwald A, Roussel M, Kroschinsky F, Lindemann W, Dreger P, Viardot A, Milpied N, Gisselbrecht C, Wulf G, Gyan E, Gaulard P, Bay JO, Glass B, Poeschel V, Damaj G, Sibon D, Delmer A, Bilger K, Banos A, Haenel M, Dreyling M, Metzner B, Keller U, Braulke F, Friedrichs B, Nickelsen M, Altmann B, Tournilhac O. A randomized phase 3 trial of autologous vs allogeneic transplantation as part of first-line therapy in poor-risk peripheral T-NHL. Blood. 2021 May 13;137(19):2646-2656. doi: 10.1182/blood.2020008825. PMID 33512419
- [Background] Tournilhac O, Altmann B, Friedrichs B, Bouabdallah K, Leclerc M, Cartron G, Turlure P, Reimer P, Wagner-Drouet E, Sanhes L, Houot R, Roussel M, Kroschinsky F, Dreger P, Viardot A, de Leval L, Rosenwald A, Gaulard P, Wulf G, Villate A, Latiere C, Elmaagacli A, Glass B, Poeschel V, Damaj G, Sibon D, Durot E, Bilger K, Banos A, Haenel M, Dreyling M, Keller U, Tiab M, Drenou B, Cornillon J, Nguyen S, Robin M, Nickelsen M, Trumper L, Lenz G, Ziepert M, Schmitz N; French Lymphoma Study Association (LYSA), the Societe Francophone de greffe de moelle et Therapie Cellulaire (SFGM-TC), and the German Lymphoma Alliance (GLA). Long-Term Follow-Up of the Prospective Randomized AATT Study (Autologous or Allogeneic Transplantation in Patients With Peripheral T-Cell Lymphoma). J Clin Oncol. 2024 Nov 10;42(32):3788-3794. doi: 10.1200/JCO.24.00554. Epub 2024 Sep 13. PMID 39270145